CLINICAL TRIAL: NCT02698150
Title: Evaluation of Remote Monitoring in Patients With Functional Mitral Regurgitation Undergoing Transcatheter Mitral Valve Edge-to-edge Repair With the Mitraclip System
Brief Title: Remote Monitoring of Patients With Functional Mitral Regurgitation Undergoing Mitraclip Transcatheter Repair
Acronym: HERMES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Ferrarotto Alessi (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Davide Capodanno, Professor, Azienda Ospedaliero, Ferrarotto Alessi
Other Study IDs: HERMES
Record Dates: First submitted 2016-02-26; First posted 2016-03-03 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Mitral Regurgitation; Heart Failure
Keywords: Mitral regurgitation; Mitraclip; Remote monitoring; Wearables
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Remote monitoring: Active group of patients undergoing daily remote monitoring using sensors and wearables
  Interventions: Device: HERMES tablet
- Control: Control group of patients undergoing standard follow up wth no remote monitoring

INTERVENTIONS:
Device: HERMES tablet — Tablet, sensors and wearables for daily collection of clinical data
  Groups: Remote monitoring

SUMMARY:
HERMES is a pilot study which aims at exploring the impact of remote monitoring in patients with severe functional mitral regurgitation undergoing transcatheter mitral valve edge-to-edge repair with the Mitraclip system.

DETAILED DESCRIPTION:
The scope of the HERMES study is to investigate whether the information obtained by remote monitoring in patients with severe functional mitral regurgitation who have undergone transcatheter mitral valve edge-to-edge repair with the Mitraclip system may have the potential to guide treatment decisions at follow-up visits, and improve the quality of life. Candidates to the Mitraclip procedure on optimal medical therapy will be offered the opportunity to participate to the study by bringing home a tablet and a series of sensors and wearables to collect daily information on blood pressure, oxygen saturation, weight variation, heart rate, symptoms and compliance to therapy. These variables will be blinded, stored by the tablet and downloaded by the core institution at follow-up visits. Clinicians will be encouraged to use these data to guide their decisions, personalizing drug therapies and follow-up schedules to the individual patient's need. Patients that during the run-in phase (from enrollment to 30+-7 days) will have used the tablet for >66% of the days will undergo the Mitraclip procedure and continue to keep the tablet for up to 12 months (active group). Patients that during the run-in phase (from enrollment to 30+-7 days) will have not used the tablet for >66% of the days, will continue the study as a control group. Predefined clinical follow up assessments for collection of study endpoints will be at 1 month post Mitraclip, 6 months post Mitraclip and 12 months post Mitraclip. Quality of life, assessed by means of the SF36v2 questionnaire, will be assessed at enrollment, pre Mitraclip, at 1 month after Mitraclip and at 12 months after Mitraclip. A series of secondary endpoints, including 6MWT assessments and consumption of resources will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic while on optimal medical therapy (NYHA Class III-IV)
* Mitral regurgitation of functional etiology
* Suitable Mitraclip candidate
* Life expectancy >12 months

Exclusion Criteria:

* Mitral regurgitation of primary etiology
* Refusal to sign the informed consent
* Dementia or neurological disorders that prevent the proper use of the tablet
* Inability to use the tablet, the sensors and/or the wearables, even with the assistance of family members
* Expected non-compliance with follow-up visits
* End-stage chronic kidney disease on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe mitral regurgitation of functional etiology undergoing transcatheter mitral valve edge-to-edge repair with the Mitraclip system
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life @ 12 months | 12 months
  Quality of life assessed with the SF36v2 questionnaire at 12 months post Mitraclip implant

SECONDARY OUTCOMES:
Quality of life @ baseline | Baseline (1 month before Mitraclip implant)
  Quality of life assessed with the SF36v2 questionnaire at 1 month before Mitraclip implant
Quality of life @ index procedure (end of the run-in phase) | pre Mitraclip implant
  Quality of life assessed with the SF36v2 questionnaire at the time of the Mitraclip procedure
Quality of life @ 1 month | 1 month after Mitraclip implant
  Quality of life assessed with the SF36v2 questionnaire at 1 month after Mitraclip implant

OTHER OUTCOMES:
6MWT (6-minute walking test) | Baseline
6MWT (6-minute walking test) | 1 month after Mitraclip implant
6MWT (6-minute walking test) | 6 months after Mitraclip implant
6MWT (6-minute walking test) | 12 months after Mitraclip implant

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tamburino, Professor, Study Chair — Ferrarotto Hospital, University of Catania; Carmelo Grasso, MD, Principal Investigator — Ferrarotto Hospital, University of Catania; Davide Capodanno, MD, PhD, Principal Investigator — Ferrarotto Hospital, University of Catania
Locations (1):
- Ferrarotto Hospital, Catania, Italy

IPD SHARING:
Plan to Share IPD: No